CLINICAL TRIAL: NCT04730999
Title: A Phase II, Single Arm Study of CarbopLatin Plus Etoposide With Bevacizumab and Atezolizumab in Patients With exTEnded-disease Small-cell Lung Cancer (SCLC)
Brief Title: Efficacy and Safety Study of a New Therapeutic Strategy in the Treatment of Extended-Disease Small-Cell Lung Cancer
Acronym: CeLEBrATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Roche Pharma, Italy (Unknown); YGHEA, CRO Division of Ecol Studio spa (Industry); Dr. Luca Boni U.O. Epidemiologia Clinica, IRCCS Ospedale Policlinico San Martino - IST NORD CBA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-01-2019; 2019-003798-25 (EudraCT Number)
Record Dates: First submitted 2020-12-21; First posted 2021-01-29 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin; Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Induction phase (6 cycles, 21 days duration): carboplatin, etoposide, bevacizumab and atezolizumab.
  Maintenance phase (12 cycles, 21 days duration): bevacizumab and atezolizumab
  Interventions: Drug: Etoposide; Drug: Carboplatin; Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Etoposide — Induction phase: 100 mg/sqm on days 1-3, for a maximum of 6 cycles (each one of 21 days duration). Intravenous administration. Treatment will continue until progression of disease, unacceptable toxicity, patient refusal.
Drug: Carboplatin — Induction phase: AUC 5 on day 1 for a maximum of 6 cycles (each one of 21 days duration). Intravenous administration. Treatment will continue until progression of disease, unacceptable toxicity, patient refusal.
Drug: Bevacizumab — Induction phase: 7.5 mg/kg on day 1, for a maximum of 6 cycles (each one of 21 days duration). Intravenous administration.
  Maintenance phase: 7.5 mg/kg on day 1, for a maximum of 12 cycles (each one of 21 days duration). Intravenous administration.
  In both phases, the treatment will continue until progression of disease, unacceptable toxicity, patient refusal.
Drug: Atezolizumab — Induction phase: flat dosing of 1200 mg on day 1, for a maximum of 6 cycles ( each one of 21 days duration). Intravenous administration.
  Maintenance phase: flat dosing of 1200 mg on day 1, for a maximum of 12 cycles (each one of 21 days duration). Intravenous administration.
  In both phases, the treatment will continue until progression of disease, unacceptable toxicity, patient refusal, loss of clinical benefit.

SUMMARY:
Small cell lung cancer (SCLC) is an aggressive type of neuroendocrine tumor with the majority of patients (about 60-70%) being diagnosed with metastatic disease and with a median survival ranging from 7 to 12 months. Combination chemotherapy (CT), namely a platinum and etoposide-based regimen, represents the cornerstone of treatment for extended disease (ED) SCLC. Despite this the duration of response is short and nearly all patients develop disease relapse or progression. The recent approval of atezolizumab in combination with carboplatin and etoposide as first line in patients with ED SCLC is surely a step forward in the understanding the molecular landscape and treatment of this complex tumor, but new therapeutic approaches need to be explored.

This trial aims to assess the efficacy in terms of 1 year survival a new therapeutic strategy that combines to the standard CT (carboplatin and etoposide), two drugs indicated in the tratment of several types of tumors: bevacizumab and atezolizomab.

The treatment will start with an induction phase during which eligible patients will receive, by intravenous way, a combination of the above mentioned drugs according to a specific administration regimen. This phase will last about 18 weeks. Therafter the treatment will proceed with a maintenence phase lasting for a maximum of 54 weeks during which the patients will receive only atezolizumab and bevacizumab, by intravenous way, according to a specific administration regimen. Treatment will be discontnued in case of disease progression, unacceptable toxicity, patient refusal or loss of clinical benefit (for atezolizumab). During the study period the patients will undergo to periodic visits and laboratory, radiologic assessments to monitor the efficacy and the safety of the ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological documented small cell lung cancer (SCLC) or poorly differentiated (G3) neuroendocrine carcinoma of the lung
* Extensive stage disease (disease which cannot be encompassed in a single radiation portal including pleural dissemination and supraclavicular node metastasis)
* No prior chemotherapy or treatment with another systemic anti-cancer agent (Note: Patients who have received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of at least 6 months since last chemotherapy, radiotherapy or chemoradiotherapy cycle from diagnosis of extended-disease SCLC)
* No need for concomitant chest irradiation
* Males or females, age ≥18 years
* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Adequate hepatic and renal functions [i.e. total bilirubin < 1.5 times the ULN; - AST and ALT < 3.0 times the ULN (AST and ALT < 5.0 x ULN is acceptable if the liver has tumor involvement); Albumin≥ 25 g/L (2.5 g/dL); serum creatinine ≤1.5 times the ULN or creatinine clearance, calculated according to the formula of Cockcroft and Gault > 60 ml/min; urine dipstick for proteinuria <2+. If urine dipstick is >2+, 24-hour urine must demonstrate ≤ 1 g of protein in 24 hours]
* Adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1500/µL, hemoglobin ≥9 g/dL (5.58 mmol/L), and platelets ≥100,000/µL.
* Adequate coagulation function as defined by International Normalized Ratio (INR) ≤1.5 and a partial thromboplastin time (PTT) (PTT/aPTT) ≤ 1.5 x upper limits of normal [ULN]. Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). If receiving warfarin, the patient must have an INR ≤3.0. For heparin and LMWH there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
* Negative HIV test at screening with respect of any applicable law and the indication of Atezolizumab use.
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. Please note: The HBV DNA test will be performed only for patients who have a positive total HBcAb test
* Negative hepatitis C virus (HCV) antibody test at screening.
* Female patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to first dose of protocol therapy.
* Male patients who are sexually active must use effective contraception during treatment with chemotherapy and for at least 6 months after the final dose of chemotherapy to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 6 months after the last dose of atezolizumab or bevacizumab. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
* Ability to comply with the study protocol, in the investigator's judgment
* Written informed consent

Exclusion Criteria:

* The patient has experienced any Grade 3-4 gastrointestinal bleeding within 3 months prior to first dose of protocol therapy.
* The patient has a history of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy.
* Symptomatic brain metastases or spinal cord compression (CT or MRI of the head is required within 4 weeks prior to registration) requiring immediate radiotherapy for palliation. Asymptomatic patients with treated or untreated CNS lesions are eligible, provided that all of the following criteria are met:

A. Presence outside the CNS of measurable disease per RECIST v1.1 B. No history of intracranial hemorrhage, spinal cord hemorrhage or heorrhagic intracranial lesions C. No stereotactic radiotherapy or whole brain radiotherapy within 14 days prior to initiation of study treatment or neurosurgical resection within 28 days prior to initiation of study treatment D. Concurrent therapy of corticosteroids ≤ 10 mg of oral prednisone or equivalent and/or anticonvulsant therapy at a stable dose E. Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla or spinal cord) F. No evidence of interim progression between completion of CNS directed therapy (if administered) and initiation of study treatment

* History of leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., Pleurocath) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected calcium > ULN)
* Active tubercolosis
* Significant traumatic injury or radiotherapy involving an extensive field within the last 4 weeks prior to first dose of study treatment or anticipation of the need for major surgery during study treatment. Palliative radiotherapy to a limited field is allowed if concluded at least 2 weeks prior enrolment.
* The patient experienced hemoptysis (defined ≥ one-half teaspoon of bright red blood per episode) within 2 months prior to first dose of protocol therapy or with radiographic evidence of intratumor cavitation.
* Other malignancies (previous or current), except for adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, localized prostate cancer surgically treated with curative intent or ductal carcinoma in situ treated surgically treated with curative intent or if previous malignancy was more than 5 years prior and there are no signs or symptoms of recurrence
* The patient has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy.
* The patient has uncontrolled or poorly-controlled hypertension (>150 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management. Anti-hypertensive therapy to achieve these parameters is allowable.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to registration
* The patient has a prior history of gastrointestinal or non-gastrointestinal fistula as well as gastrointestinal perforation (within 6 months of first dose of protocol therapy) or risk factors for perforation.
* The patient has a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy.
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgery (including open biopsy) within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to the first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
* Prior allogeneic stem cell or solid organ transplantation
* Patients with any underlying medical condition that might be aggravated by treatment or which cannot be controlled i.e. patients with active serious infection, diabetes mellitus, pericardial effusion.
* Concomitant treatment with any other anti-cancer drug
* Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to starting study treatment
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
* Active, known or suspected autoimmune disease. Subjects with hypothyroidism only requiring hormone replacement, type I diabetes or autoimmune skin disorders not requiring systemic treatments are permitted to enroll.
* Patient has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Active infection requiring therapy.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), Hepatitis B (HBV) or Hepatitis C (HCV)
* History of idiopathic pulmonary fibrosis, including pneumonitis, drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, CD137 agonists.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment.
* Any condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of registration. Steroid doses of ≤ 10 mg daily prednisone equivalent are permitted.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* History of allergies or hypersensitivity to any study drugs or study drug components.
* The patient is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Interval between the date of enrolment and the date of death from any cause, up to a maximum of 25 months.
  Percentage of patients surviving 1 year after study treatment end

SECONDARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events [Safety and Tolerability] | Interval between the date of enrolment and the date of death from any cause, up to a maximum of 15 months
  Frequency of adverse events. Severity of adverse events measured according to NCI Common Toxicity Criteria Adverse Event (CTCAE), version 5.0.
Overall Response Rate (ORR) | Interval between the date of enrolment and the date of death from any cause, up to a maximum of 13 months.
  The sum of complete response (CR) + partial response (PR). Tumor responses will be evaluated according to standard RECIST 1.1 criteria. Patients with no tumor assessment after baseline will be classified as non-responders.
Progression-Free Survival (PFS) | Interval between the date of enrolment and the date of progressive disease, or death, up to a maximum of 13 months.
  The time of survival without progression of disease confirmed according to to standard RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, Dr, Principal Investigator — S. Orsola-Malpighi University Hospital - Dept. Oncology-Haematology; Karim Rihawi, Dr, Study Chair — S. Orsola-Malpighi University Hospital - Dept. Oncology-Haematology
Locations (14):
- Italy (14):
  - UOC di Oncologia Medica - AOU Policlinico S. Orsola Malpighi, Bologna
  - UOC Oncologia Medica - PO A.Perino - ASL di Brindisi, Brindisi
  - UOC Medicina Oncologica - Ospedale di Carpi - Azienda USL di Modena, Carpi
  - UO di Oncologia - Istituti Ospitalieri di Cremona - ASST Di Cremona, Cremona
  - UOC Oncologia Medica - AO S. Croce e Carle di Cuneo, Cuneo
  - UOC di Oncologia Ematologia - AOU di Ferrara, Ferrara
  - UOC Oncologia Medica 1 - AOU Careggi, Florence
  - Oncologia medica - Policlinico San Martino, Genova
  - UOC Oncologia Medica - Azienda ULSS9 Veneto, Legnago
  - Dip. Oncologia-Ematologia - UO Oncologia - AOU Policlinico di Modena, Modena
  - UOC Oncologia Medica - AORN "A. Cardarelli", Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - UOC di Oncologia Medica - AOU di Parma, Parma
  - Dipartimento di Oncologia ASUIUD, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brattstrom D, Bergqvist M, Hesselius P, Larsson A, Wagenius G, Brodin O. Serum VEGF and bFGF adds prognostic information in patients with normal platelet counts when sampled before, during and after treatment for locally advanced non-small cell lung cancer. Lung Cancer. 2004 Jan;43(1):55-62. doi: 10.1016/j.lungcan.2003.07.007. PMID 14698537
- [Background] Giatromanolaki A. Prognostic role of angiogenesis in non-small cell lung cancer. Anticancer Res. 2001 Nov-Dec;21(6B):4373-82. PMID 11908693
- [Background] Souhami RL, Spiro SG, Rudd RM, Ruiz de Elvira MC, James LE, Gower NH, Lamont A, Harper PG. Five-day oral etoposide treatment for advanced small-cell lung cancer: randomized comparison with intravenous chemotherapy. J Natl Cancer Inst. 1997 Apr 16;89(8):577-80. doi: 10.1093/jnci/89.8.577. PMID 9106647
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Evans WK, Shepherd FA, Feld R, Osoba D, Dang P, Deboer G. VP-16 and cisplatin as first-line therapy for small-cell lung cancer. J Clin Oncol. 1985 Nov;3(11):1471-7. doi: 10.1200/JCO.1985.3.11.1471. PMID 2997406
- [Background] Goldie JH, Coldman AJ. A mathematic model for relating the drug sensitivity of tumors to their spontaneous mutation rate. Cancer Treat Rep. 1979 Nov-Dec;63(11-12):1727-33. PMID 526911
- [Background] Roth BJ, Johnson DH, Einhorn LH, Schacter LP, Cherng NC, Cohen HJ, Crawford J, Randolph JA, Goodlow JL, Broun GO, et al. Randomized study of cyclophosphamide, doxorubicin, and vincristine versus etoposide and cisplatin versus alternation of these two regimens in extensive small-cell lung cancer: a phase III trial of the Southeastern Cancer Study Group. J Clin Oncol. 1992 Feb;10(2):282-91. doi: 10.1200/JCO.1992.10.2.282. PMID 1310103
- [Background] Jain RK. Normalizing tumor vasculature with anti-angiogenic therapy: a new paradigm for combination therapy. Nat Med. 2001 Sep;7(9):987-9. doi: 10.1038/nm0901-987. No abstract available. PMID 11533692
- [Background] Reck M, Crino L. Advances in anti-VEGF and anti-EGFR therapy for advanced non-small cell lung cancer. Lung Cancer. 2009 Jan;63(1):1-9. doi: 10.1016/j.lungcan.2008.05.015. Epub 2008 Jun 25. PMID 18579254
- [Background] Horn L, Dahlberg SE, Sandler AB, Dowlati A, Moore DF, Murren JR, Schiller JH. Phase II study of cisplatin plus etoposide and bevacizumab for previously untreated, extensive-stage small-cell lung cancer: Eastern Cooperative Oncology Group Study E3501. J Clin Oncol. 2009 Dec 10;27(35):6006-11. doi: 10.1200/JCO.2009.23.7545. Epub 2009 Oct 13. PMID 19826110
- [Background] Ready NE, Dudek AZ, Pang HH, Hodgson LD, Graziano SL, Green MR, Vokes EE. Cisplatin, irinotecan, and bevacizumab for untreated extensive-stage small-cell lung cancer: CALGB 30306, a phase II study. J Clin Oncol. 2011 Nov 20;29(33):4436-41. doi: 10.1200/JCO.2011.35.6923. Epub 2011 Oct 3. PMID 21969504
- [Background] Spigel DR, Greco FA, Zubkus JD, Murphy PB, Saez RA, Farley C, Yardley DA, Burris HA 3rd, Hainsworth JD. Phase II trial of irinotecan, carboplatin, and bevacizumab in the treatment of patients with extensive-stage small-cell lung cancer. J Thorac Oncol. 2009 Dec;4(12):1555-60. doi: 10.1097/JTO.0b013e3181bbc540. PMID 19875975
- [Background] Spigel DR, Townley PM, Waterhouse DM, Fang L, Adiguzel I, Huang JE, Karlin DA, Faoro L, Scappaticci FA, Socinski MA. Randomized phase II study of bevacizumab in combination with chemotherapy in previously untreated extensive-stage small-cell lung cancer: results from the SALUTE trial. J Clin Oncol. 2011 Jun 1;29(16):2215-22. doi: 10.1200/JCO.2010.29.3423. Epub 2011 Apr 18. PMID 21502556
- [Background] Pujol JL, Morin F, Zalcman G; IFCT. Reply to the letter to the editor 'Flaws in the trial design of IFCT-0802' by Gyawali et al. Ann Oncol. 2015 Oct;26(10):2199. doi: 10.1093/annonc/mdv292. Epub 2015 Aug 7. No abstract available. PMID 26254441
- [Background] Tiseo M, Boni L, Ambrosio F, Camerini A, Vitale MG, Baldini E, Cinieri S, Zanelli F, Defraia E, Passalacqua R, Crino L, Dazzi C, Tibaldi C, Turolla GM, D'Alessandro V, Zilembo N, Riccardi F, Ardizzoni A; Gruppo Oncologico Italiano di Ricerca Clinica (GOIRC). Italian multicenter phase III randomized study of cisplatin-etoposide with or without bevacizumab as first-line treatment in extensive stage small cell lung cancer: treatment rationale and protocol design of the GOIRC-AIFA FARM6PMFJM trial. Clin Lung Cancer. 2015 Jan;16(1):67-70. doi: 10.1016/j.cllc.2014.09.001. Epub 2014 Sep 28. PMID 25450879
- [Background] Tiseo M, Boni L, Ambrosio F, Camerini A, Baldini E, Cinieri S, Brighenti M, Zanelli F, Defraia E, Chiari R, Dazzi C, Tibaldi C, Turolla GM, D'Alessandro V, Zilembo N, Trolese AR, Grossi F, Riccardi F, Ardizzoni A. Italian, Multicenter, Phase III, Randomized Study of Cisplatin Plus Etoposide With or Without Bevacizumab as First-Line Treatment in Extensive-Disease Small-Cell Lung Cancer: The GOIRC-AIFA FARM6PMFJM Trial. J Clin Oncol. 2017 Apr 20;35(12):1281-1287. doi: 10.1200/JCO.2016.69.4844. Epub 2017 Jan 30. PMID 28135143
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Reck M, Heigener D, Reinmuth N. Immunotherapy for small-cell lung cancer: emerging evidence. Future Oncol. 2016 Apr;12(7):931-43. doi: 10.2217/fon-2015-0012. Epub 2016 Feb 17. PMID 26882955
- [Background] Ott PA, Elez E, Hiret S, Kim DW, Morosky A, Saraf S, Piperdi B, Mehnert JM. Pembrolizumab in Patients With Extensive-Stage Small-Cell Lung Cancer: Results From the Phase Ib KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 1;35(34):3823-3829. doi: 10.1200/JCO.2017.72.5069. Epub 2017 Aug 16. PMID 28813164
- [Background] Antonia SJ, Lopez-Martin JA, Bendell J, Ott PA, Taylor M, Eder JP, Jager D, Pietanza MC, Le DT, de Braud F, Morse MA, Ascierto PA, Horn L, Amin A, Pillai RN, Evans J, Chau I, Bono P, Atmaca A, Sharma P, Harbison CT, Lin CS, Christensen O, Calvo E. Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2016 Jul;17(7):883-895. doi: 10.1016/S1470-2045(16)30098-5. Epub 2016 Jun 4. PMID 27269741
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, Sengupta S, Frank I, Parker AS, Zincke H, Blute ML, Sebo TJ, Cheville JC, Kwon ED. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006 Apr 1;66(7):3381-5. doi: 10.1158/0008-5472.CAN-05-4303. PMID 16585157
- [Background] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Background] Okazaki T, Honjo T. PD-1 and PD-1 ligands: from discovery to clinical application. Int Immunol. 2007 Jul;19(7):813-24. doi: 10.1093/intimm/dxm057. Epub 2007 Jul 2. PMID 17606980
- [Background] Hino R, Kabashima K, Kato Y, Yagi H, Nakamura M, Honjo T, Okazaki T, Tokura Y. Tumor cell expression of programmed cell death-1 ligand 1 is a prognostic factor for malignant melanoma. Cancer. 2010 Apr 1;116(7):1757-66. doi: 10.1002/cncr.24899. PMID 20143437
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Socinski MA, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Kelsch C, Lee A, Coleman S, Deng Y, Shen Y, Kowanetz M, Lopez-Chavez A, Sandler A, Reck M; IMpower150 Study Group. Atezolizumab for First-Line Treatment of Metastatic Nonsquamous NSCLC. N Engl J Med. 2018 Jun 14;378(24):2288-2301. doi: 10.1056/NEJMoa1716948. Epub 2018 Jun 4. PMID 29863955
- [Background] Huang Y, Chen X, Dikov MM, Novitskiy SV, Mosse CA, Yang L, Carbone DP. Distinct roles of VEGFR-1 and VEGFR-2 in the aberrant hematopoiesis associated with elevated levels of VEGF. Blood. 2007 Jul 15;110(2):624-31. doi: 10.1182/blood-2007-01-065714. Epub 2007 Mar 21. PMID 17376891
- [Background] Shrimali RK, Yu Z, Theoret MR, Chinnasamy D, Restifo NP, Rosenberg SA. Antiangiogenic agents can increase lymphocyte infiltration into tumor and enhance the effectiveness of adoptive immunotherapy of cancer. Cancer Res. 2010 Aug 1;70(15):6171-80. doi: 10.1158/0008-5472.CAN-10-0153. Epub 2010 Jul 14. PMID 20631075
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Bouzin C, Feron O. Targeting tumor stroma and exploiting mature tumor vasculature to improve anti-cancer drug delivery. Drug Resist Updat. 2007 Jun;10(3):109-20. doi: 10.1016/j.drup.2007.03.001. Epub 2007 Apr 23. PMID 17452119
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Nishino M, Giobbie-Hurder A, Gargano M, Suda M, Ramaiya NH, Hodi FS. Developing a common language for tumor response to immunotherapy: immune-related response criteria using unidimensional measurements. Clin Cancer Res. 2013 Jul 15;19(14):3936-43. doi: 10.1158/1078-0432.CCR-13-0895. Epub 2013 Jun 6. PMID 23743568